CLINICAL TRIAL: NCT05971602
Title: A Phase 2b/c, Multi-Arm, 2-Stage, Duration Randomized Trial of the Efficacy and Safety of Two to Four Months Treatment With Regimens Containing Bedaquiline, OPC-167832, and Sutezolid, Plus Either Pretomanid or Delamanid, in Adults With Pulmonary Tuberculosis
Brief Title: Efficacy and Safety Evaluation of Two to Four Months of Treatment With the Combination Regimens of DBOS and PBOS in Adults With Pulmonary Tuberculosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Data generated in the Gates MRI-TBD06-201 trial do not support the investigational regimens being able to achieve the trial objective of identifying a new regimen to treat tuberculosis in 3 months or less.
Sponsor: Gates Medical Research Institute (Other)
Collaborators: Global Alliance for TB Drug Development (Other); Janssen Pharmaceuticals (Industry); Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Gates MRI-TBD06-201
Record Dates: First submitted 2023-06-14; First posted 2023-08-02 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Pulmonary Tuberculosis
Keywords: Delamanid, Bedaquiline, OPC-167832, and Sutezolid (DBOS); Pretomanid, Bedaquiline, OPC-167832, and Sutezolid (PBOS); Drug sensitive tuberculosis; Rifampicin-resistant tuberculosis (RR-TB); Multi-drug resistant tuberculosis (MDR-TB)
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis, Multidrug-Resistant | interventions — OPC-67683; bedaquiline; PNU-100480; pretomanid; Isoniazid; Rifampin; Pyrazinamide; Ethambutol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (10):
- Stage 1: Arm 1: DS-TB Participants receiving DBOS for 4 months (17 Weeks) (Experimental)
  Interventions: Drug: Delamanid, Bedaquiline, OPC-167832, and Sutezolid (DBOS)
- Stage 1: Arm 2: DS-TB Participants receiving PBOS for 4 months (17 Weeks) (Experimental)
  Interventions: Drug: Pretomanid, Bedaquiline, OPC-167832, and Sutezolid (PBOS)
- Stage 1: Arm 3: DS-TB Participants receiving 2HRZE/4HR for 6 months (26 weeks) (Experimental): Isoniazid (H), Rifampicin (R), Pyrazinamide (Z), Ethambutol (E) - refers to standard regimen of 8 weeks of HRZE followed by 18 weeks of HR (2HRZE/4HR)
  Interventions: Drug: Isoniazid, Rifampicin, Pyrazinamide, Ethambutol (HRZE); Drug: Isoniazid and Rifampicin (HR)
- Stage 2: Arm 1: DS-TB Participants receiving XBOS for 2 months (9 Weeks) (Experimental): Pretomanid or Delamanid, Bedaquiline, OPC-167832, and Sutezolid (Regimen from Stage 1 that advances to Stage 2 [XBOS])
  Interventions: Drug: Pretomanid or Delamanid, Bedaquiline, OPC-167832, and Sutezolid (XBOS)
- Stage 2: Arm 2: DS-TB Participants receiving XBOS for 2.5 months (11 Weeks) (Experimental)
  Interventions: Drug: Pretomanid or Delamanid, Bedaquiline, OPC-167832, and Sutezolid (XBOS)
- Stage 2: Arm 3: DS-TB Participants receiving XBOS for 3 months (13 Weeks) (Experimental)
  Interventions: Drug: Pretomanid or Delamanid, Bedaquiline, OPC-167832, and Sutezolid (XBOS)
- Stage 2: Arm 4: DS-TB Participants receiving XBOS for 3.5 months (15 Weeks) (Experimental)
  Interventions: Drug: Pretomanid or Delamanid, Bedaquiline, OPC-167832, and Sutezolid (XBOS)
- Stage 2: Arm 5: DS-TB Participants receiving XBOS for 4 months (17 Weeks) (Experimental)
  Interventions: Drug: Pretomanid or Delamanid, Bedaquiline, OPC-167832, and Sutezolid (XBOS)
- Stage 2: Arm 6: DS-TB Participants receiving 2HRZE/4HR for 6 months (26 Weeks) (Experimental)
  Interventions: Drug: Isoniazid, Rifampicin, Pyrazinamide, Ethambutol (HRZE); Drug: Isoniazid and Rifampicin (HR)
- Observational cohort: RR/MDR-TB Participants receiving XBOS for 4 months (17 Weeks) (Experimental)
  Interventions: Drug: Pretomanid or Delamanid, Bedaquiline, OPC-167832, and Sutezolid (XBOS)

INTERVENTIONS:
Drug: Delamanid, Bedaquiline, OPC-167832, and Sutezolid (DBOS) — D- 300 milligram (mg) once daily (QD) for treatment duration; B- 400 mg QD for 2 weeks, 200 mg thrice weekly for remaining treatment weeks; O- 30 mg QD for treatment duration and S- 1200 mg QD for treatment duration
  Arms: Stage 1: Arm 1: DS-TB Participants receiving DBOS for 4 months (17 Weeks)
Drug: Pretomanid, Bedaquiline, OPC-167832, and Sutezolid (PBOS) — P- 200 mg QD for treatment duration; B- 400 mg QD for 2 weeks, 200 mg thrice weekly for remaining treatment weeks; O- 30 mg QD for treatment duration and S- 1200 mg QD for treatment duration
  Arms: Stage 1: Arm 2: DS-TB Participants receiving PBOS for 4 months (17 Weeks)
Drug: Isoniazid, Rifampicin, Pyrazinamide, Ethambutol (HRZE) — Fixed dose combination (FDC) of 75 mg of isoniazid, 150 mg of rifampicin, 400 mg of pyrazinamide, and 275 mg of ethambutol (HRZE) (Standard of Care [SOC]). All the doses administered will be weight-based.
  Arms: Stage 1: Arm 3: DS-TB Participants receiving 2HRZE/4HR for 6 months (26 weeks); Stage 2: Arm 6: DS-TB Participants receiving 2HRZE/4HR for 6 months (26 Weeks)
Drug: Pretomanid or Delamanid, Bedaquiline, OPC-167832, and Sutezolid (XBOS) — X - Pretomanid 200 mg QD for treatment duration OR Delamanid 300 mg QD for treatment duration; B - 400 mg QD for 2 weeks, 200 mg thrice weekly for remaining treatment weeks; O- 30 mg QD for treatment duration and S-1200 mg QD for treatment duration
  Arms: Observational cohort: RR/MDR-TB Participants receiving XBOS for 4 months (17 Weeks); Stage 2: Arm 1: DS-TB Participants receiving XBOS for 2 months (9 Weeks); Stage 2: Arm 2: DS-TB Participants receiving XBOS for 2.5 months (11 Weeks); Stage 2: Arm 3: DS-TB Participants receiving XBOS for 3 months (13 Weeks); Stage 2: Arm 4: DS-TB Participants receiving XBOS for 3.5 months (15 Weeks); Stage 2: Arm 5: DS-TB Participants receiving XBOS for 4 months (17 Weeks)
Drug: Isoniazid and Rifampicin (HR) — Fixed dose combination (FDC) of 75 mg of isoniazid and 150 mg of rifampicin (HR) (Standard of Care [SOC]). All the doses administered will be weight-based.
  Arms: Stage 1: Arm 3: DS-TB Participants receiving 2HRZE/4HR for 6 months (26 weeks); Stage 2: Arm 6: DS-TB Participants receiving 2HRZE/4HR for 6 months (26 Weeks)

SUMMARY:
This multicenter, two-stage, open-label, randomized trial will aim to assess the efficacy, safety, optimal duration, and pharmacokinetics (PK) of Delamanid, Bedaquiline, OPC-167832, and Sutezolid (DBOS) and Pretomanid, Bedaquiline, OPC-167832, and Sutezolid (PBOS) in adult participants with drug sensitive tuberculosis (DS-TB) and rifampicin or multi-drug resistant TB (RR/MDR-TB).

ELIGIBILITY:
Inclusion Criteria:

For Stage 1:

* Able to provide written, informed consent prior to initiation of any trial-related procedures or treatments, and able, in the opinion of the Investigator, to comply with all the requirements of the trial.
* Male or female participants between 18 and 65 years of age (inclusive) at the screening visit.
* Body weight ≥35.0 kilograms (kg) and body mass index (BMI) ≥16.0 at the screening visit.
* Newly diagnosed within the past 8 weeks prior to informed consent, untreated (≤4 days of treatment), drug-susceptible pulmonary TB, as defined by all of the following:

  1. Confirmation of Mtb infection: Mtb positivity on a molecular test (eg, Xpert Ultra, Hain Line probe assay [LPA]) conducted on a sputum specimen for trial screening.
  2. Evidence of non-paucibacillary disease: ≥1+ sputum smear positivity for acid-fast bacilli using fluorescent microscopy, as defined by the International Union Against Tuberculosis and Lung Disease (IUATLD)/World Health Organization (WHO) scale, OR a Xpert Ultra semi-quantitative result of 'medium' or 'high' on the sputum specimen for trial screening.
  3. Drug-susceptible TB: Isoniazid and rifampicin resistance not detected, as determined by a molecular test (eg, Hain LPA, Xpert Ultra, Xpert MTB/Extensively Drug Resistant [XDR]) conducted on a sputum specimen for trial screening.
  4. Clinical signs and/or symptoms consistent with active TB in the opinion of the Investigator.
  5. Chest radiograph consistent with active TB in the opinion of the Investigator. Note, the Investigator is permitted, but not required, to incorporate a radiologist's interpretation into their assessment of a participant's chest radiograph.
* Able to spontaneously produce sputum.
* Female participants of childbearing potential (FOCBP) must agree to use 2 approved methods of contraception with their male sexual partners or abstain from heterosexual intercourse throughout their participation in the trial.
* Male participants must agree to use an approved method of contraception with their female sexual partners of childbearing potential or abstain from heterosexual intercourse throughout their participation in the trial.

For Stage 2:

• Newly diagnosed within the past 8 weeks of informed consent, untreated (≤4 days of treatment), drug-susceptible or rifampicin-/multi-drug resistant pulmonary TB, as defined by all of the following:

1. Confirmation of Mtb infection: Mtb positivity on a molecular test (eg, Xpert Ultra, Hain LPA) conducted on a screening sputum specimen.
2. Evidence of non-paucibacillary disease: ≥1+ sputum smear positivity for acid-fast bacilli using fluorescent microscopy, as defined on the IUATLD/WHO scale, OR Xpert Ultra semi-quantitative result of 'medium' or 'high' on the sputum specimen for trial screening.
3. Resistance pattern:

i. For DS TB arm, isoniazid and rifampicin resistance not detected on a molecular test (eg, Hain LPA, Xpert Ultra, Xpert MTB/XDR) conducted on a screening sputum specimen, OR

ii. For RR/MDR TB arm, either rifampicin resistance (RR TB) OR rifampicin and isoniazid resistance (MDR TB) detected on a molecular test (eg, Hain LPA, Xpert Ultra, Xpert MTB/XDR) conducted on a screening sputum specimen.

• Participants with RR or MDR TB must also have fluoroquinolone resistance not detected, as determined by a molecular test (eg, Hain LPA second line, Xpert MTB/XDR) performed on the sputum specimen for trial screening.

d) Clinical signs and/or symptoms consistent with active TB in the opinion of the Investigator.

e) Chest radiograph consistent with active TB in the opinion of the Investigator.

The other inclusion criteria remain the same for Stage 2.

Exclusion Criteria:

* Suspected or documented extra-thoracic TB. Confirmed or suspected lymph node TB is not considered exclusionary. The presence of a pleural effusion considered not clinically significant together with pulmonary TB is not exclusionary.
* Known, or suspected of having, resistance to a rifamycin, isoniazid, ethambutol, pyrazinamide, delamanid, pretomanid, bedaquiline, linezolid, tedizolid, or sutezolid either confirmed by the laboratory, or based on epidemiological history, such as a known source case with said resistance.
* Received any prior treatment for active Mtb disease (>4 days) within the past 1 year of informed consent.
* Received any treatment with a fluoroquinolone active against Mtb (ie, levofloxacin, moxifloxacin, ciprofloxacin) or an aminoglycoside for more than 14 days within the 3 months prior to informed consent even if the medication was given for a different indication than TB treatment.
* Any known prior exposure to delamanid, pretomanid, bedaquiline, OPC-167832, or any oxazolidinone (linezolid, tedizolid, delpazolid, or sutezolid).
* Evidence of an active clinically significant/uncontrolled metabolic, gastrointestinal, neurological (including peripheral neuropathy), psychiatric, endocrine (including uncontrolled diabetes), hematologic, ophthalmologic (particularly optic neuritis), or liver disease; active malignancy; or other medical co-morbidity considered significant enough by the Investigator that the participant should not enter the trial.
* Significant history of, or current clinically relevant cardiovascular disorder, such as heart failure, coronary artery disease, uncontrolled hypertension, arrhythmia, tachyarrhythmia, prolonged QT syndrome, or presence of symptom(s) strongly suggestive of such a problem, such as exertional chest pressure/pain or unexplained syncope.
* Significant history of, or current evidence of an active clinically significant/poorly controlled pulmonary disease, such as asthma, Chronic obstructive Pulmonary disease (COPD), silicosis, or lung fibrosis (other than TB), considered as severe by the Investigator. In particular, any underlying pulmonary condition that could significantly interfere with the assessment of X-ray images, interpretation of sputum findings, or otherwise compromise the participant's participation in the trial is exclusionary based on the Investigator's judgement. Clinically significant post-Coronavirus disease-2019 (COVID-19) pulmonary sequelae should be considered exclusionary.
* If HIV-infected, having any of the following present:

  1. Not on antiretroviral treatment at time of screening or taking antiretroviral treatment for <3 months prior to screening, OR
  2. Cluster of differentiation (CD)4+ T-cell count <200 cells/microliter (μL) during the screening period, OR
  3. HIV viral load >200 copies/milliliter (mL) during the screening period, OR
  4. Evidence of a currently active opportunistic malignancy or infection related to HIV other than TB that requires treatment with a prohibited concomitant medication (oral candidiasis is not exclusionary) OR
  5. HIV-infected participants enrolling at a trial site in Peru will not be eligible due to the requirement for longer TB treatment courses than the standard 6-month HRZE regimen for patients with HIV/TB co-infection as per the Peruvian national TB treatment guidelines.
* If female, currently pregnant or breastfeeding, OR having a positive serum or urine pregnancy test during the screening period, OR planning to become pregnant within the 12-month period after the screening period.
* Current significant drug and/or alcohol abuse that is likely to result in poor adherence to trial requirements or that would pose a risk to the participant's wellbeing during the trial.
* Karnofsky Performance Status scale score at screening of <60.
* Having a disease or condition where the use of delamanid, pretomanid, bedaquiline, OPC-167832, sutezolid, rifampicin, isoniazid, pyrazinamide, or ethambutol is contraindicated.
* Positive Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Polymerase chain reaction (PCR) result on nasopharyngeal sample taken during screening. Prior history of COVID-19/SARS-CoV-2 infection is not exclusionary if SARS-CoV-2 PCR performed on screening sample is negative.
* Any of the following laboratory results during screening:

  1. Estimated creatinine clearance <60 mL/minute
  2. Alanine transaminase (ALT) or aspartate transaminase (AST) >2.5 × upper limit of normal of the clinical laboratory reference range
  3. Total bilirubin >2x upper limit of normal of the clinical laboratory reference range, at screening
  4. Hemoglobin <8.0 grams per deciliter (g/dL)
  5. Platelet count <100 x 10^9/liter (L)
  6. White blood cell count <2.0 x 10^9/L
  7. Screening glycosylated hemoglobin (HbA1c) ≥10.0%
  8. Positive hepatitis B surface antigen
  9. Positive hepatitis C antibody.
* Moderate to severe substance use disorder according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria (substances of concern may include cocaine, amphetamines, opiates, barbiturates, benzodiazepines, or alcohol).
* A clinically significant Electrocardiogram (ECG) abnormality at screening as confirmed by a central ECG reading service. Examples of such include, but are not limited to, second- or third-degree atrioventricular block, complete right bundle branch block, left bundle branch block, QRS duration ≥120 millisecond (msec), QT interval corrected using Fridericia's formula (QTcF) interval >450 msec in males or >470 msec in females, atrial fibrillation or flutter, supraventricular tachycardia, and ventricular tachycardia or multiple multifocal premature ventricular complexes. The following ECG findings are not considered clinically significant: sinus tachycardia, mild first-degree atrioventricular block (P-R interval <0.23 sec), right or left axis deviation, incomplete right bundle branch block, and isolated left anterior fascicular block (left anterior hemiblock) in young otherwise healthy participants.
* Participants receiving any of the prohibited medications within the specified periods or who would be likely to require prohibited concomitant therapy during the trial.
* History of having taken another investigational drug within 30 days preceding trial entry or participates in another clinical study during the duration of this trial.
* Prospective approvals of protocol deviations to enrollment criteria, also known as protocol waivers or exemptions, are not permitted.
* Participants with baseline culture results (defined as collected during screening period through up to Week 1) that are all negative for growth of Mtb will not be included in efficacy analyses. DS-TB participants whose baseline phenotypic DST results demonstrate resistance to isoniazid and/or rifampicin will not be included in efficacy analyses. Their treatment will be modified accordingly based on their resistance profile, relevant local/national guidelines, and the participant's interest to continue in the trial after discussion with the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2023-07-26 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
Stage 1: Percentage of participants with DS-TB reporting severe Adverse events (AEs) (≥ Grade 3) and/or Serious adverse events (SAEs), by treatment group | Up to Week 19 for DBOS and PBOS; up to Week 28 for 2HRZE/4HR
Stage 1: Percentage of participants with pulmonary DS-TB with unfavorable outcome, by treatment group | At Week 17 for DBOS and PBOS; at Week 26 for 2HRZE/4HR
  Participants that experience one or more of the following events following randomization will be categorized as having an unfavorable outcome status: Absence of microbiological cure (positive sputum culture); Death from any cause; Permanent discontinuation of trial treatment before the end of the assigned treatment duration ; Extension of TB treatment by the Investigator more than 5 days beyond the end of the assigned treatment duration for any reason; Positive culture for Mtb at last visit excluding documented TB re-infection with a different Mtb strain than Baseline.
Stage 2: Percentage of participants with DS-TB reporting severe AEs (≥ Grade 3) and/or SAEs, by treatment group | Up to Week 19 for XBOS treatment groups; up to Week 28 for 2HRZE/4HR
Stage 2: Percentage of participants with pulmonary DS-TB reporting unfavorable outcome, by treatment group | At 12 months post-randomization
  Participants that experience one or more of the following events following randomization will be categorized as having an unfavorable outcome status: Absence of microbiological cure (positive sputum culture); Death from any cause; Permanent discontinuation of trial treatment before the end of the assigned treatment duration; Extension of TB treatment by the Investigator more than 5 days beyond the end of the assigned treatment duration for any reason; Re-start of TB treatment by the Investigator during the post-treatment follow-up period excluding documented TB re-infection with a different Mtb strain than Baseline; Positive culture for Mtb at last visit excluding documented TB re-infection with a different Mtb strain than Baseline.

SECONDARY OUTCOMES:
Stage 1: Percentage of participants reporting all-cause trial treatment discontinuation, by treatment group | Through 12 months post-randomization
Stage 1: Percentage of participants reporting severe AEs (≥ Grade 3) and/or SAEs, by treatment group | Through 12 months post-randomization
Stage 1: Percentage of participants with pulmonary DS-TB and Human immunodeficiency virus (HIV) co-infection reporting severe AEs (≥ Grade 3) and/or SAEs, by treatment group | Up to Week 19 for DBOS and PBOS; up to Week 28 for 2HRZE/4HR
Stage 1: Percentage of participants with pulmonary DS-TB and HIV co-infection reporting severe AEs (≥ Grade 3) and/or SAEs, by treatment group | Through 12 months post-randomization
Stage 1: Percentage of participants with pulmonary DS-TB and HIV co-infection reporting all-cause trial treatment discontinuation, by treatment group | Through 12 months post-randomization
Stage 1: Percentage of participants with pulmonary DS-TB reporting unfavorable outcome, by treatment group | At 12 months post-randomization
  Participants that experience one or more of the following events following randomization will be categorized as having an unfavorable outcome status: Absence of microbiological cure (positive sputum culture); Death from any cause; Permanent discontinuation of trial treatment before the end of the assigned treatment duration; Extension of TB treatment by the Investigator more than 5 days beyond the end of the assigned treatment duration for any reason; Re-start of TB treatment by the Investigator during the post-treatment follow-up period excluding documented TB re-infection with a different Mtb strain than Baseline; Positive culture for Mtb at last visit excluding documented TB re-infection with a different Mtb strain than Baseline.
Stage 1: Percentage of participants with DS-TB and HIV co-infection reporting unfavorable outcome, by treatment group | At Week 17 for DBOS and PBOS; at Week 26 for 2HRZE/4HR
  Participants that experience one or more of the following events following randomization will be categorized as having an unfavorable outcome status: Absence of microbiological cure (positive sputum culture); Death from any cause; Permanent discontinuation of trial treatment before the end of the assigned treatment duration; Extension of TB treatment by the Investigator more than 5 days beyond the end of the assigned treatment duration for any reason; Re-start of TB treatment by the Investigator during the post-treatment follow-up period excluding documented TB re-infection with a different Mtb strain than Baseline; Positive culture for Mtb at last visit excluding documented TB re-infection with a different Mtb strain than Baseline.
Stage 1: Percentage of participants reporting unfavorable outcome, by treatment group | At 6 months post-randomization
  Participants that experience one or more of the following events following randomization will be categorized as having an unfavorable outcome status: Absence of microbiological cure (positive sputum culture); Death from any cause; Permanent discontinuation of trial treatment before the end of the assigned treatment duration; Extension of TB treatment by the Investigator more than 5 days beyond the end of the assigned treatment duration for any reason; Re-start of TB treatment by the Investigator during the post-treatment follow-up period excluding documented TB re-infection with a different Mtb strain than Baseline; Positive culture for Mtb at last visit excluding documented TB re-infection with a different Mtb strain than Baseline.
Stage 1: Time to sustained sputum culture conversion to negative for Mtb growth in Mycobacteria Growth Indicator Tube (MGIT) culture in participants receiving combination of DBOS and PBOS relative to 2HRZE/4HR | Up to Week 28
  Hazard ratio for time to sustained sputum culture conversion to negative will be assessed
Stage 1: Mean change from Baseline in sputum MGIT culture time to detection (TTD) in participants receiving combination of DBOS and PBOS relative to 2HRZE/4HR | Baseline and at Weeks 4, 8, 9, 13, and 17
  Mean change from Baseline in sputum MGIT culture time to detection (TTD) will be assessed
Stage 1: Percentage of participants with sustained sputum culture conversion in MGIT culture through Week 26, by treatment group | Through Week 26 post-randomization
Stage 1: Time to sustained sputum culture conversion to negative in solid culture, by treatment group | Up to Week 19 for DBOS and PBOS; up to Week 28 for 2HRZE/4HR
Stage 1: Percentage of participants with sustained sputum culture conversion in solid culture, by treatment group | Up to Week 19 for DBOS and PBOS; up to Week 28 for 2HRZE/4HR
Stage 1: Percentage of participants developing resistance against each drug | Up to 12 months post-randomization
Stage 1: Change from Baseline in minimum inhibitory concentration (MIC) for delamanid, pretomanid, bedaquiline, OPC-167832, and sutezolid drugs | Up to 12 months post-randomization
Stage 1: Geometric mean concentration of DBOS in participants with pulmonary DS-TB | Pre-dose, post-dose at Weeks 1, 2, 4, 6, 9, 11, 13, 15, 17, 19, 21, 23, 26 and at Months 9, 12
Stage 1: Geometric mean concentration of PBOS in participants with pulmonary DS-TB | Pre-dose, post-dose at Weeks 1, 2, 4, 6, 9, 11, 13, 15, 17, 19, 21, 23, 26 and at Months 9, 12
Stage 1: Geometric mean concentration of DBOS in participants with DS-TB and HIV co-infection | Pre-dose, post-dose at Weeks 1, 2, 4, 6, 9, 11, 13, 15, 17, 19, 21, 23, 26 and at Months 9, 12
Stage 1: Geometric mean concentration of PBOS in participants with DS-TB and HIV co-infection | Pre-dose, post-dose at Weeks 1, 2, 4, 6, 9, 11, 13, 15, 17, 19, 21, 23, 26 and at Months 9, 12
Stage 1: Geometric coefficient of variation of DBOS in participants with pulmonary DS-TB | Pre-dose, post-dose at Weeks 1, 2, 4, 6, 9, 11, 13, 15, 17, 19, 21, 23, 26 and at Months 9, 12
Stage 1: Geometric coefficient of variation of PBOS in participants with pulmonary DS-TB | Pre-dose, post-dose at Weeks 1, 2, 4, 6, 9, 11, 13, 15, 17, 19, 21, 23, 26 and at Months 9, 12
Stage 1: Geometric coefficient of variation of DBOS in participants with DS-TB and HIV co-infection | Pre-dose, post-dose at Weeks 1, 2, 4, 6, 9, 11, 13, 15, 17, 19, 21, 23, 26 and at Months 9, 12
Stage 1: Geometric coefficient of variation of PBOS in participants with DS-TB and HIV co-infection | Pre-dose, post-dose at Weeks 1, 2, 4, 6, 9, 11, 13, 15, 17, 19, 21, 23, 26 and at Months 9, 12
Stage 2: Percentage of participants with DS-TB receiving XBOS reporting all-cause trial treatment discontinuation | Week 9 through 17
Stage 2: Percentage of participants with DS-TB receiving 2HRZE/4HR reporting all-cause trial treatment discontinuation | Up to week 26
Stage 2: Percentage of participants with DS-TB reporting Severe AEs (≥ Grade 3) and/or SAEs, by treatment group | Through 12 months post-randomization
Stage 2: Percentage of participants with pulmonary DS-TB and HIV co-infection reporting severe AEs (≥ Grade 3) and/or SAEs, by treatment group | Up to Week 11, Week 13, Week 15, Week 17, and Week 19 for XBOS treatment groups; up to Week 28 for 2HRZE/4HR
Stage 2: Percentage of participants with pulmonary DS-TB and HIV co-infection reporting severe AEs (≥ Grade 3) and/or SAEs, by treatment group | Through 12 months post-randomization
Stage 2: Percentage of participants with pulmonary DS-TB and HIV co-infection reporting all-cause trial treatment discontinuation, by treatment group | Up to Week 9, Week 11, Week 13, Week 15, and Week 17 for XBOS treatment groups; up to Week 26 for 2HRZE/4HR
Stage 2: Percentage of participants with RR/MDR-TB reporting severe AEs (≥ Grade 3) and/or SAEs in participants who receive XBOS for four months | Up to 19 weeks
Stage 2: Percentage of participants with RR/MDR-TB reporting severe AEs (≥ Grade 3) and/or SAEs in participants who receive XBOS for four months | Through 12 months post-randomization
Stage 2: Percentage of participants with RR/MDR-TB reporting all-cause trial treatment discontinuation in participants who receive XBOS for four months | Up to 17 weeks
Stage 2: Percentage of participants with pulmonary DS-TB reporting unfavorable outcome, by treatment group | Week 9, Week 11, Week 13, Week 15, and Week 17 for XBOS treatment groups; at Week 26 for 2HRZE/4HR
  Participants that experience one or more of the following events following randomization will be categorized as having an unfavorable outcome status: Absence of microbiological cure (positive sputum culture); Death from any cause; Permanent discontinuation of trial treatment before the end of the assigned treatment duration ; Extension of TB treatment by the Investigator more than 5 days beyond the end of the assigned treatment duration for any reason; Positive culture for Mtb at last visit excluding documented TB re-infection with a different Mtb strain than Baseline.
Stage 2: Percentage of participants with pulmonary DS-TB and HIV co-infection reporting unfavorable outcome, by treatment group | Through 12 months post-randomization
  Participants that experience one or more of the following events following randomization will be categorized as having an unfavorable outcome status: Absence of microbiological cure (positive sputum culture); Death from any cause; Permanent discontinuation of trial treatment before the end of the assigned treatment duration; Extension of TB treatment by the Investigator more than 5 days beyond the end of the assigned treatment duration for any reason; Re-start of TB treatment by the Investigator during the post-treatment follow-up period excluding documented TB re-infection with a different Mtb strain than Baseline; Positive culture for Mtb at last visit excluding documented TB re-infection with a different Mtb strain than Baseline.
Stage 2: Percentage of participants reporting unfavorable outcome, by treatment group | At 6 months post-treatment after randomized duration of treatment
  Participants that experience one or more of the following events following randomization will be categorized as having an unfavorable outcome status: Absence of microbiological cure (positive sputum culture); Death from any cause; Permanent discontinuation of trial treatment before the end of the assigned treatment duration; Extension of TB treatment by the Investigator more than 5 days beyond the end of the assigned treatment duration for any reason; Re-start of TB treatment by the Investigator during the post-treatment follow-up period excluding documented TB re-infection with a different Mtb strain than Baseline; Positive culture for Mtb at last visit excluding documented TB re-infection with a different Mtb strain than Baseline.
Stage 2: Time to sustained sputum culture conversion to negative for Mtb growth in MGIT culture in participants receiving combination of XBOS relative to 2HRZE/4HR | Up to Week 28
Stage 2: Mean change from Baseline in sputum MGIT culture TTD in participants receiving combination of XBOS relative to 2HRZE/4HR | Baseline and at Weeks 4, 8, 9, 11, 13, 15, and 17
Stage 2: Percentage of participants with sustained sputum culture conversion to negative at Week 8 and end of treatment, by treatment group | At Week 8 for all treatment groups; at Week 9, Week 11, Week 13, Week 15, and Week 17 for all XBOS treatment groups; at Week 26 for 2HRZE/4HR
Stage 2: Time to sustained sputum culture conversion to negative in solid culture in participants receiving combination of XBOS relative to 2HRZE/4HR | Up to Week 28
Stage 2: Percentage of participants with sustained sputum culture conversion in solid culture, by treatment group | Up to Week 11, Week 13, Week 15, Week 17, and Week 19 for XBOS treatment groups; up to Week 28 for 2HRZE/4HR
Stage 2: Percentage of participants with sustained sputum culture conversion to negative by each treatment group | Up to Week 28
Stage 2: Percentage of participants developing resistance against each drug | Up to 12 months post-randomization
Stage 2: Change from Baseline in MIC for delamanid, pretomanid, bedaquiline, OPC-167832, and sutezolid drugs | Up to 12 months post-randomization
Stage 2: Geometric mean concentration of XBOS in participants with pulmonary DS-TB and RR/MDR-TB | Pre-dose, post-dose at Weeks 1, 2, 4, 6, 9, 11, 13, 15, 17, 19, 21, 23, 26 and at Months 9, 12
Stage 2: Geometric mean concentration of XBOS in participants with DS-TB and HIV co-infection | Pre-dose, post-dose at Weeks 1, 2, 4, 6, 9, 11, 13, 15, 17, 19, 21, 23, 26 and at Months 9, 12
Stage 2: Geometric coefficient of variation of XBOS in participants with pulmonary DS-TB and RR/MDR-TB | Pre-dose, post-dose at Weeks 1, 2, 4, 6, 9, 11, 13, 15, 17, 19, 21, 23, 26 and at Months 9, 12
Stage 2: Geometric coefficient of variation of XBOS in participants with DS-TB and HIV co-infection | Pre-dose, post-dose at Weeks 1, 2, 4, 6, 9, 11, 13, 15, 17, 19, 21, 23, 26 and at Months 9, 12

CONTACTS AND LOCATIONS:
Overall Officials: Gates MRI, Study Director — Gates Medical Research Institute
Locations (13):
- Philippines (3):
  - Tropical Disease Foundation, Makati
  - Lung Center of the Philippines, Quezon City
  - Silang Specialist Medical Center, Silang
- South Africa (10):
  - Bio-Medical Research Institute; Faculty of Medicine and Health Sciences, Stellenbosch University; Tygerberg Medical Campus, Cape Town
  - TASK - Central (Brooklyn), Cape Town
  - UCT (Cape Town); General Medicine & Global Health (GMGH); Hatter Heart Research Institute, Cape Town
  - UCT South African Tuberculosis Vaccine Initiative (SATVI), Cape Town
  - University of Cape Town (UCT) Lung Institute, Cape Town
  - CHRU - Durban, Durban
  - Synergy Biomed Research Institute, East London
  - Clinical HIV Research Unit (CHRU) - Johannesburg, Johannesburg
  - The Aurum Institute (Tembisa CRS), Johannesburg
  - Perinatal HIV Research Unit (PHRU), Klerksdorp

IPD SHARING:
Plan to Share IPD: Yes